CLINICAL TRIAL: NCT00397956
Title: An Open-Label, Single-Arm, Non-Comparative Study to Evaluate the Efficacy, Tolerability & Convenience of Invanz(TM) (Ertapenem Sodium) In the Treatment of Community-Acquired Sepsis in Adults
Brief Title: To Evaluate the Treatment Effect of an Anti-Infective Agent for Complicated Infections (0826-053)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0826-053; 2006_047
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Ertapenem; Duration of Therapy

INTERVENTIONS:
Drug: MK0826, ertapenem sodium / Duration of Treatment: 14 Days

SUMMARY:
To collect clinical response data with the use of ertapenem in community acquired sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 years of age or older
* Patients present with at least two of the following signs and symptom:
* fever (temperature> 38c or < 36c)
* heart rate > 90 beats/min)
* respiratory rate> 20 breaths/min)
* high white blood cell count > 12,000/ul or >10% bands)

Exclusion Criteria:

* Patient has a history of allergy or hypersensitivity (anaphylaxis) or serious adverse reaction to ertapenem or any carbapenem
* Patient has a poor chance of survival for more than 14 days.
* Patient has an apache ii score > 15 (see attachment 3.
* Patient has an infection caused by pathogens resistant to ertapenem
* The patient requires antibiotics other than ertapenem (such as: glycopeptides, macrolides or antifungal agents)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms of infection on days 3, 4, 7 and 14 during treatment

SECONDARY OUTCOMES:
Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC